CLINICAL TRIAL: NCT07092137
Title: Nano-crystalline Megestrol Acetate for Anorexia-Cachexia in Advanced Lung Cancer: A Randomized, Double-Blind, Multicenter Study
Brief Title: Nano-crystalline Megestrol Acetate for Anorexia-Cachexia Syndrome in Advanced Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Vice President of the First Affiliated Hospital of Guangzhou Medical University, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGA-25-0701
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Cachexia-Anorexia Syndrome
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nanocrystalline megestrol acetate+immunochemotherapy (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension
- Nanocrystalline megestrol acetate placebo+immunochemotherapy (Placebo Comparator)
  Interventions: Other: Nano-crystalline Megestrol Acetate Oral Suspension placebo

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nano-crystalline Megestrol Acetate+PD-(L)1 inhibitor (Q3W, until PD) + chemotherapy (based on guidelines)
  Arms: Nanocrystalline megestrol acetate+immunochemotherapy
Other: Nano-crystalline Megestrol Acetate Oral Suspension placebo — Nano-crystalline Megestrol Acetate placebo+PD-(L)1 inhibitor (Q3W, until PD) + chemotherapy (based on guidelines)
  Arms: Nanocrystalline megestrol acetate placebo+immunochemotherapy

SUMMARY:
Patients with advanced lung cancer are a high-risk population for cancer-related anorexia-cachexia syndrome (CACS). Meanwhile, the adverse reactions of chemotherapy and immunotherapy potentially exacerbate the occurrence and progression of CACS. CACS seriously affects the quality of life of patients with advanced lung cancer, significantly shortens the overall survival (OS) and progression-free survival (PFS), forming a vicious cycle. A number of previous studies have shown that combined supportive therapies such as megestrol acetate during chemotherapy or concurrent chemoradiotherapy for advanced tumor patients is a clinically meaningful and feasible treatment model in clinical practice. However, the efficacy and optimal treatment timing of combination with current first-line immunochemotherapy regimens remain unclear. Although mechanistic studies have shown that anti-cachexia therapy may synergistically enhance the efficacy of immunotherapy, relevant clinical research evidence is lacking.

Therefore, this study hypothesizes that the combination of first-line immunochemotherapy regimen and nano-crystalline megestrol acetate can improve the clinical benefits of patients with advanced lung cancer. It is planned to enroll patients with advanced lung cancer who present with anorexia-cachexia, and administer nano-crystalline megestrol acetate intervention (nano-crystalline megestrol acetate or its placebo control) during first-line immunochemotherapy. The changes in body weight relative to the baseline, as well as the impact on survival benefits and quality of life of patients, will be detected. In China, megestrol acetate is mainly available in two dosage forms: oral suspension and dispersible tablets. The oral suspension of megestrol acetate adopts nano-crystal technology (referred to as nano-crystalline megestrol acetate), which reduces the particle size of megestrol acetate and improves bioavailability. Previous randomized controlled studies have shown that it is superior to non-nano-crystal dosage forms in improving body weight.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible for study enrollment:

1. Inclusion criteria for advanced lung cancer:

   1. Patients with histologically or cytologically confirmed locally advanced (Stage ⅢC) or metastatic (Stage IV) non-small cell lung cancer (NSCLC) that cannot be completely resected surgically or treated with radical chemoradiotherapy, according to the 8th edition of the TNM staging classification for lung cancer by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer Classification.
   2. Patients with histologically or cytologically confirmed small cell lung cancer (SCLC) and diagnosed as extensive-stage SCLC based on the 8th edition of AJCC staging or the Veterans Administration Lung Group (VALG) criteria (excluding mixed small cell lung cancer).
   3. Subjects who have not received prior systemic chemotherapy for metastatic disease. Subjects who received adjuvant/neoadjuvant chemotherapy or radical concurrent/sequential chemoradiotherapy with curative intent for non-metastatic disease are eligible if disease progression occurs >6 months after the end of the last treatment.
   4. At least one measurable tumor lesion according to RECIST v1.1.
2. Criteria for pre-cachexia or cachexia stage:

   1. Pre-cachexia diagnostic criteria (all three must be met):

      * Unintentional weight loss ≤5% in the past 6 months;

        ② Systemic inflammation (CRP >5 mg/L);

        ③ Decreased appetite (FAACT-A/CS 12 score ≤37).
   2. Fearon diagnostic criteria for cachexia stage (any one of the following combined with decreased appetite [FAACT-A/CS 12 score ≤37] or systemic inflammation [CRP >5 mg/L]):

      * Unintentional weight loss >5% in the past 6 months; ② Weight loss >2% when BMI <18.5 kg/m².
3. General inclusion requirements:

   1. Good compliance and signed informed consent form.
   2. Age 18-75 years, regardless of gender.
   3. ECOG performance status 0-2.
   4. Life expectancy ≥6 months.
   5. Good organ function:

      • Hematological: Neutrophils ≥1.5×10⁹/L, hemoglobin ≥9 g/dL, platelets ≥100×10⁹/L.

      • Liver function: Bilirubin ≤1.5×ULN (patients with known Gilbert disease and serum bilirubin ≤3×ULN are eligible); AST and ALT ≤2.5×ULN (if liver metastasis is present, AST and ALT ≤5×ULN); alkaline phosphatase ≤3×ULN (if liver or bone metastasis is present, ALP ≤5×ULN); albumin ≥3 g/dL.
      * Coagulation function: International normalized ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (aPTT) ≤1.5×ULN.
      * Renal function: Creatinine clearance rate ≥60 mL/min (calculated by Cockcroft-Gault formula).
      * Urine protein ≤1+ or 24-hour urine protein <1.0 g.
      * Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%.
   6. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 3 days before the first drug administration (if the urine test is inconclusive, a serum test is required, with the serum result as the standard). If a female patient of childbearing potential has sexual activity with an unsterilized male partner, she must use an acceptable contraceptive method from screening and agree to continue contraception for 120 days after the last administration of the study drug. Whether to discontinue contraception after this period should be discussed with the investigator. Male patients who are not sterilized and have sexual activity with female partners of childbearing potential must use effective contraception from screening to 120 days after the last administration. Whether to discontinue contraception after this period should be discussed with the investigator.

Exclusion Criteria:

* (1) Cancer-specific exclusion criteria:

  a) Active or untreated CNS metastases (e.g., brain or leptomeningeal metastases) confirmed by CT or magnetic resonance (MRI) evaluation during screening and prior imaging. Patients who have received treatment for brain or leptomeningeal metastases, have been stable for ≥2 months, and have discontinued systemic hormonal therapy (>10 mg/d prednisone or equivalent) >4 weeks before randomization may participate.

  b) Uncontrolled tumor-related pain. c) Thromboembolic disease, ascites, or lower limb edema within the past 6 months.

  d) History of malignant tumors other than lung cancer within 5 years before randomization, except for malignancies with negligible risk of metastasis or death [e.g., expected 5-year overall survival rate >90%] and expected to be cured after treatment, such as appropriately treated cervical in situ carcinoma, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery.

  e) Unresolved toxicity from prior antitumor therapy, defined as failure to recover to NCI CTCAE v5.0 grade 0 or 1 (except alopecia) or to the levels specified in the inclusion/exclusion criteria.

  (2) General medical exclusion criteria:
  1. Women who are pregnant, lactating, or planning to become pregnant during the study.
  2. Patients with hepatitis B (known HBsAg-positive and HBV DNA ≥1000 cps/ml or 200 IU/ml or ≥ the upper limit of normal at each study center) or hepatitis C:

     ● For patients with a history of HBV infection, HBV DNA testing must be performed, and they are eligible only if HBV DNA is negative (HBV DNA <1000 cps/ml or 200 IU/ml or below the upper limit of normal).
     * Among patients with positive HCV antibody, only those with negative HCV RNA by polymerase chain reaction (PCR) may participate.
  3. Patients with positive human immunodeficiency virus (HIV) test results.
  4. Receipt of major surgery (excluding diagnostic surgery) within 28 days before randomization, or expected to undergo major surgery during the study.
  5. Significant cardiovascular diseases, such as heart disease defined by the New York Heart Association (class II or higher), myocardial infarction within 3 months before randomization, unstable arrhythmia, unstable angina, cerebrovascular accident, or transient ischemic attack. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must receive the optimal stable treatment regimen as determined by their attending physician, with consultation from a cardiologist if necessary.
  6. Severe infection within 4 weeks before the first drug administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks before the first drug administration (excluding antiviral therapy for hepatitis B or C).

     (3) Medication-related exclusion criteria:

  <!-- -->

  1. Any condition affecting gastrointestinal absorption, such as dysphagia, malabsorption, uncontrollable vomiting; patients with difficulty in food intake or requiring enteral or parenteral nutrition support; anorexia nervosa, anorexia due to mental illness, or difficulty in eating due to pain.
  2. Current or planned use of other appetite or weight-increasing medications, such as adrenal corticosteroids (except short-term dexamethasone use during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
  3. Patients with Cushing's syndrome, adrenal or pituitary insufficiency; poorly controlled diabetes; current hypertension with systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite oral antihypertensive treatment.
  4. History of esophageal-gastric varices, severe ulcers, gastrointestinal perforation and/or fistula, gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months before the first drug administration.
  5. Known allergy to any component of the study drug.
  6. Other circumstances deemed unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with a body weight increase of >5% relative to the baseline. | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
appetite | From enrollment to the end of treatment at 12 week
  The proportion of participants with a better appetite >5% relative to the baseline. Participants report a score on a scale FAACT-A/CS 12，with 4 higher scores mean a better outcome.
QOL | From enrollment to the end of treatment at 12 week
  Participants report a score on a scale EORTC QLQ-C30.
Anxiety and depression | From enrollment to the end of treatment at 12 week
  Participants report a score on a scale HADS
PFS in 6 months and 12 months | From enrollment to the end of treatment at 6 months and 12 months
Treatment compliance ( relative dose intensity, RDI) | From enrollment to the end of treatment at 12 weeks
  Relative Dose Intensity (RDI): The ratio of the actual administered dose intensity to the standard planned dose intensity, usually expressed as a percentage (%).
L3-SMI | From enrollment to the end of treatment at 12 weeks
  The Hounsfield unit (HU) limits used for assessing skeletal muscle mass ranged from -29 to +150 HU. The muscle area was normalised for height, resulting in a ratio (cm2/m2) known as the L3 skeletal mass index (L3 SMI).
Inflammatory indicators (CRP, IL-1, IL-6, TNF-α, etc.) | From enrollment to the end of treatment at 12 weeks
Nutritional indicators (prealbumin, albumin, hemoglobin) | From enrollment to the end of treatment at 12 weeks
ACTH、VIP、SSTR | From enrollment to the end of treatment at 12 weeks

IPD SHARING:
Plan to Share IPD: Yes